CLINICAL TRIAL: NCT03799211
Title: Adherence to and Beliefs on Recommendations for Behavioral Treatment for Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-00937
Record Dates: First submitted 2018-12-31; First posted 2019-01-10 (Actual); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Motivational Interviewing; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental)
  Interventions: Behavioral: Motivational Interviewing
- Usual Care (Active Comparator)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Motivational Interviewing — Phone call using motivational interviewing technique
  Arms: Motivational Interviewing
Behavioral: Treatment as Usual — will receive a regular study phone call after three months
  Arms: Usual Care

SUMMARY:
Migraine patients are oftentimes referred for evidence based behavioral therapies to prevent migraine. Yet, at follow-up visits, they report not seeing the behavioral therapist. This is a pilot feasibility acceptability study to assess whether motivational interviewing (MI) can be implemented in the headache center setting to help improve initiation and adherence to behavioral therapy for migraine. We will also assess patients' reasons for making/not making the appointment.

ELIGIBILITY:
Inclusion Criteria:

* Migraine diagnosis age 16+
* English speaking

Exclusion Criteria:

* Unable to read the questionnaire, no phone number

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mia Minen, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Interviewing | Usual Care
Started | 36 | 40
Completed | 32 | 27
Not Completed | 4 | 13
Not completed — Lost to Follow-up | 2 | 13
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing | Usual Care | Total
Number analyzed (Participants) | 36 | 40 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.3) | 38.1 (12.1) | 39.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 39 | 71
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 30 | 36 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 26 | 33 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 36 | 40 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Made an Appointment for Behavioral Therapy
Time Frame: 3-6 Months
Measure: Number; unit: percentage of participants
Arm/Group | Motivational Interviewing | Usual Care
Number analyzed (Participants) | 32 | 27
percentage of participants | 37.5 | 22.2

2. Secondary Outcome: Percentage of Participants Who Attended Appointments
Description: Of those who initiated behavioral therapy, percentage who attended appointments
Time Frame: 3-6 Months
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Motivational Interviewing
Number analyzed (Participants) | 27 | 32
percentage of participants | 22.2 | 21.9

3. Secondary Outcome: Percentage of Participants Who Initiated Appointments
Time Frame: Month 3-4 post-recruitment
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | Motivational Interviewing
Number analyzed (Participants) | 27 | 32
percentage of participants | 40.7 | 68.8

4. Secondary Outcome: Mean Reported Importance of Managing Migraine
Description: Reported the importance to participants of managing migraine. Importance was rated on a scale from 0 to 10, where the higher the score, the higher the importance.
Time Frame: First Follow-up Call (1 month post baseline) conducted only for the Arm/Group "Motivational Interviewing" and Last Follow-up Call (3-4 months post baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Motivational Interviewing
Number analyzed (Participants) | 27 | 32
units on a scale
  First Follow-Up Call | NA (NA) — Only one follow-up call was conducted for this arm | 9.16 (1.27)
  Last Follow-Up Call | 9.19 (1.3) | 9.22 (1.18)

5. Secondary Outcome: Mean Reported Confidence in Managing Migraines
Description: Reported confidence in participant's ability to manage migraine. Confidence was rated on a scale from 0 to 10, with the higher the score, the higher the confidence.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Motivational Interviewing
Number analyzed (Participants) | 27 | 32
score on a scale
  First Follow-Up Call | NA (NA) — Only one follow-up call was conducted for this arm | 6.26 (2.27)
  Last Follow-Up Call | 6.59 (2.26) | 6.62 (2.50)

6. Secondary Outcome: Mean Reported Confidence in Behavioral Therapy
Description: Reported confidence in behavioral therapy to help participant manage migraine. Confidence was rated on a scale from 0 to 10, where the higher the score, the higher the confidence.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Motivational Interviewing
Number analyzed (Participants) | 27 | 32
score on a scale
  First Follow-Up Call | NA (NA) — Only one follow-up call was conducted for this arm | 4.83 (2.47)
  Last Follow-Up Call | 5.35 (2.59) | 5.04 (1.95)

ADVERSE EVENTS:
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study.
Arm/Group | Motivational Interviewing | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03799211/Prot_SAP_000.pdf